CLINICAL TRIAL: NCT01487785
Title: A Phase Ib, Open-label, Multicenter, Dose-escalation, Safety and Tolerability Study of LDE225 in Combination With Gemcitabine in Patients With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Dose-escalation, and Safety Study of LDE225 and Gemcitabine in Locally Advanced or Metastatic Pancreatic Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X2103; 2010-024218-70 (EudraCT Number)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-01

CONDITIONS: Pancreatic Cancer
Keywords: metastatic pancreatic cancer; LDE225; gemcitabine; locally advanced; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

ARMS (1):
- LDE225+gemcitabine (Experimental): Increasing doses of LDE225 (from 400 mg) once a day + 1000 mg/m2 of gemcitabine on days 1, 8 and 15 of every 28 day cycle.
  Interventions: Drug: LDE225+gemcitabine

INTERVENTIONS:
Drug: LDE225+gemcitabine — Patients will receive increasing doses of LDE225 (from 400 mg), depending on the cohort they are assigned to, orally once daily and standard doses of gemcitabine (1000 mg/m2) on days 1, 8 and 15 of every 28-day cycle. Patients will receive the study treatment until they progressed, experience unacceptable toxicity, withdraw from the study, or the investigator decides it is in their best interest to discontinue the study treatment.

SUMMARY:
This phase Ib study includes two phases: dose escalation phase and safety expansion phase.

During the dose escalation phase, successive cohorts of eligible patients (minimum 3 and maximum 6 evaluable patients per cohort) will receive increasing oral doses of LDE225 administered on a continuous once daily (QD) dose in combination of gemcitabine. This phase of the study will determine the maximum tolerated dose (MTD) and/ or recommended dose for expansion (RDE) of LDE225 administered in combination with gemcitabine in locally advanced or metastatic pancreatic adenocarcinoma patients.

During the safety expansion phase, once the MTD of LDE225 is established, additional patients will be enrolled and treated at the MTD of LDE225 in combination with gemcitabine in order to further evaluate its safety, tolerability and explore the potential efficacy of the combined treatments on the patients in locally advanced or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic pancreatic adenocarcinoma that have not been previously treated or have progressed despite chemotherapy
* Performance status of 0 or 1 per WHO classification
* Adequate hematologic , renal and liver function
* Adequate blood creatine kinase value (CK < 1.5ULN)

Exclusion Criteria:

* Treatment with prior radiotherapy
* Pancreatic cancer that is potentially curable by surgery
* Women of childbearing potential unless they are using highly effective method of contraception Other protocol-defined inclusion/exclusion criteria may apply

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate and category of dose limiting toxicities (DLTs) | first 8 weeks of study treatment
  Dose limiting toxicities that occur during the first 8 weeks (56 days) of treatment with LDE225+gemcitabine. Dose limiting toxicity is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications that meets study specific criteria.

SECONDARY OUTCOMES:
Incidence rate of Adverse Events and Serious Adverse Events | at Informed Consent Form (ICF) sign off until 120 days after the last dose of study drug
  Adverse events and serious adverse events, changes in hematology and chemistry values and assessment of physical and neurological examinations, vital signs and electrocardiograms that occur during the reported period
Plasma pharmacokinetics(PK) parameters of LDE225 | baseline, week 9 of the study
  Area Under the Curve (AUC), Maximum observed plasma concentration after drug administration (Cmax), Time to reach Cmax (Tmax), etc.
Plasma pharmacokinetics (PK) of gemcitabine | Baseline, week 9 of the study
  If possible: AUC, Cmax, Tmax, Half life (T1/2), Total body clearance (CL), Apparent volume of distribution at steady state (Vss)
Antitumor efficacy of LDE225+gemcitabine | baseline, week 9 of the study
  Efficacy endpoints (Objective response rate and progression free survival) as a function of Hh target gene expression in tumor samples
Progression free survival | baseline, 8 weeks
  the effect of LDE225+gemcitabine on progression free survival. Progression Free Survival is defined as the time from date of enrollment to the date of the first documented progression, or death due to any cause, or start of new anti-cancer therapy.
Objective Response Rate | Baseline, 8 weeks
  The effect of LDE225+gemcitabine on objective response rate. Objective response rate is defined as the proportion of patients with a confirmed complete response (CR) or partial response (PR) as their best overall response per RECIST 1.0
Duration of Response | Baseline, 8 weeks
  The effect of LDE225+gemcitabine on duration of response. Duration of response is defined as the time from the first occurrence of complete response or partial response until the date of the first documented disease progression or death due to underlying cancer.
Serum tumor marker Ca 19-9 | On Day 1 of every cycle (cycle = 28 days)
  the effect of LDE225+gemcitabine on changes overtime in the serum tumor marker Ca 19-9 levels from baseline as assessed by central lab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (3):
  - Massachusetts General Hospital Dept. of Mass General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center MSKCC - SC, New York, New York
  - University of Utah / Huntsman Cancer Institute Huntsman UT, Salt Lake City, Utah
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Liverpool, United Kingdom

REFERENCES:
- See also: Results for CLDE225X2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13924